CLINICAL TRIAL: NCT05333211
Title: A Blinded, Randomized Controlled Study Investigating the Safety of Ortho-R® for Rotator Cuff Repair Compared With Standard of Care
Brief Title: Ortho-R® for Rotator Cuff Repair Compared With Standard of Care Rotator Cuff Repair Without Ortho-R®
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ChitogenX Inc (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ORT-2020-01
Record Dates: First submitted 2022-03-31; First posted 2022-04-18 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2022-06

CONDITIONS: Rotator Cuff Tears
Keywords: Shoulder Repair
MeSH Terms: conditions — Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Investigational Arm with Ortho-R/PRP (Experimental): Using a double row, Trans-osseous Equivalent Rotator Cuff Repair Technique (TOE) with Ortho-R/PRP combination
  Interventions: Drug: Ortho-R/PRP
- Control Arm Standard of Care without Ortho-R/PRP (No Intervention): Using the Trans-osseous Equivalent Rotator Cuff Repair Technique (TOE) without Ortho-R/PRP combination

INTERVENTIONS:
Drug: Ortho-R/PRP — Ortho-R® is a freeze-dried drug/biologic combination product containing a chitosan component and trehalose, a disaccharide that acts as a lyoprotectant during the lyophilization process and calcium chloride, which acts as a PRP coagulation agent.
  Arms: Investigational Arm with Ortho-R/PRP

SUMMARY:
Phase I/II, multi-center, prospective, blinded 2arm, parallel design and randomized controlled study. Assessing the Ortho-R/PRP combination and standard of care for rotator cuff repair, will be compared though 12 months.

DETAILED DESCRIPTION:
Phase I/II, multi-center, prospective, blinded 2arm, parallel design and randomized controlled study. Three subjects will be treated with the investigational arm and will service as training cases. The next 2 randomized intervention cases will be staggered by 48-96 hours and observed for adverse events. Randomized enrollment will then be initiated for all participating sites. Assessment of subjects with Ortho-R/PRP combination with be compared to subjects not randomized to Ortho-R/PRP group receiving standard of care who undergo rotator cuff repair surgery. Patients will be assessed by collecting patient-reported outcomes, MRI, incidence of rotator cuff re-tears, hematology and all adverse events. Data from pre-operative evaluation, day of surgery, and post-operative at 10 days, and 1,3, 6 and 12 months will be collected.

ELIGIBILITY:
Inclusion Criteria:

* Subject is ≥40 to ≤75 years.
* Subject has a primary symptomatic fully repairable rotator cuff tear ranging between 1.5 to 4 cm involving the supraspinatus and/or infraspinatus that is amenable to a TOE repair.
* Subject's rotator cuff tear must be repaired arthroscopically.
* Subject has failed at least 6 weeks of conservative management, from symptoms onset, of at least 2 conservative treatments including oral pain medications [including but not limited to non-narcotics, NSAIDs, acetaminophen as per labeling of the medications], chiropractic care, rest and structured physical therapy or exercise program prescribed by physical therapist, chiropractor provider or physician specifically for the treatment of rotator cuff tear injuries; or demonstrates the presence of unacceptable progressive symptoms or signs of acute functional deficit or intractable pain for which conservative care as noted above is otherwise not indicated.
* Subject has full passive movement of the arm comparable to the normal unaffected shoulder.
* If subject is female or male, and of reproductive capacity, subject must be:

  1. Actively practicing a contraception method throughout the study,
  2. Practicing abstinence,
  3. Surgically sterilized, or
  4. Postmenopausal.
* Subject agrees to not use any NSAIDs e.g., naproxen, high dose aspirin, ibuprofen, Meloxicam, Diclofenac, etc., and/or Paracetamol for 5 days prior to baseline, 1 week (7 days) prior to surgery and for 6 weeks post-surgery with the exception of low dose aspirin. In addition, subject must agree to not use these products within 5 days of each follow-up visit starting with the 3-month visit, so as not to introduce confounding factors for assessments.
* Subject is willing and able to return for protocol required follow-up visits.
* Subject is willing and able to voluntarily sign the IRB approved Informed Consent.

Exclusion Criteria:

* Subject with body mass index (BMI) ≤20 and ≥35.
* Subject has any of the following conditions in the index shoulder:

  1. Received a cortisone injection within 3 months prior to Surgery (Day 0)
  2. Loss of ligaments
  3. Known neuromuscular or neurovascular compromise.
  4. Deltoid deficiency (defect, tear, palsy).
  5. Samilson-Prieto Grade > 2 for osteoarthritis of glenohumeral joint.
  6. Subject has a Goutallier Grade ≥3 fatty infiltration.
  7. History within the past 5 years of anterior or posterior shoulder subluxation or dislocation as determined by history, examination or radiographic findings.
* Subject has a partial rotator cuff tear.
* Subject's condition is bilateral and rotator cuff repair is scheduled or is to be scheduled over the course of this study for the contralateral shoulder.
* Subject has had prior or current involvement of the subscapularis or teres minor.
* Subject requires concurrent fracture repair or reconstruction of the index shoulder.
* Subject has a known allergy to shellfish.
* Subject has any of the following conditions:

  1. thrombocytopenia,
  2. anemia,
  3. platelet dysfunction syndrome,
  4. hemodynamic instability or septicemia,
* Subject has had a recent fever or illness.
* Subject has prior rotator cuff tendon repair, or ≥2 prior corticosteroid injections in the index shoulder.
* Subject has an underlying metabolic bone disease (e.g., Paget's disease, fibrous dysplasia, osteoporosis).
* Subject is at a higher risk for post-surgical bleeding (e.g., bleeding disorders; taking anticoagulants except low dose aspirin) or post-surgical infection (e.g., taking immunosuppressants; has a severe infection or recent use of systemic steroids).
* Subject has a known collagen disorder, including systemic lupus erythematous (SLE), rheumatoid arthritis (RA), polymyositis, scleroderma, ankylosing spondylitis, dermatomyositis, osteogenesis imperfecta or the inherited disorders of Sjogren, Larsen, Raynaud, Ehlers-Danlos or Marfan syndrome.
* Subject has any disease, condition or surgery which in the opinion of investigator might impair healing, such as an active malignancy, history of metastatic malignancy, inflammatory or auto-immune based joint disease.
* Subject has evidence of a systemic infection, infection of the index shoulder or infection of the shoulder joint or overlying tissue such as septic arthritis, overlying cellulitis, or adjacent osteomyelitis.
* Subject has history of peripheral or central vascular disease, renal dysfunction, liver disease, COPD, uncontrolled asthma, coagulopathies, cancers aside from basal cell carcinomas, uncontrolled neurological conditions, ongoing HIV, hepatitis B or C, active tuberculosis, recurrent infections, uncontrolled cardiac arrhythmias, or mental/emotional disorders that are not well controlled.
* Subject has diagnosed musculoskeletal cancer, or any other diagnosed cancer not on long term remission (e.g., at least 5 years or negative biopsy at last exam) except basal cell carcinoma.
* Subject who demonstrates any clinically significant abnormality* for any of the following hematology testing within 30 days (± 2days) of enrollment:

  1. Complete blood count with differential
  2. Blood chemistry [comprehensive metabolic panel including aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (ALP), bilirubin, creatinine, and CRP), coagulation profile (including international normalized ration (INR), prothrombin time (PT), activated partial thromboplastin time (APTT)]
  3. Thrombin Time (TT) and
  4. Fibrinogen (FIB).
* Subject who demonstrates any clinically significant abnormality* for any of the following vital signs within 30 days (± 2days) of enrollment:

  1. Systolic BP > 160 mmHg or < 90 mmHg
  2. Pulse > 100 bpm or < 60 bpm
  3. Respiratory Rate > 25 or < 10
  4. O2 saturation < 90% on Room Air.
* Subject with any mental or psychological disorder that would impair their decisional capability.
* Subject has uncontrolled, defined as HB A1c of > 8.0%, or insulin-dependent diabetes.
* Subject with a documented history of substance abuse within six months of treatment.
* Subject has known claustrophobia and/or contraindications to MR imaging.
* Subjects with any clinically significant finding that, in the investigator's judgment, would place the subject at health risk, impact the study, or affect the completion of the study.
* Subject has any medical problem that precludes the subject from undergoing elective surgery.
* Subjects who are participating concurrently in another clinical study or have participated in a clinical study within 30 days of surgery (Day 0) or intend to during the course of the study.
* Subject is pregnant.
* Subject taking systemic steroids (excluding inhalers) and/or auto-immune suppressor drugs within 3 months prior to surgery (Day 0) or who are at risk of needing systemic steroids, such as for asthma.
* Subjects who are currently involved in any injury litigation relating to the index shoulder.
* Subjects with stiffness due to Adhesive Capsulitis.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2022-07-26 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
Complications | Day of surgery
  Assess adverse events and serious adverse events and patient safety
Complications | post-operative 10 days
  Assess adverse events and serious adverse events and patient safety
Complications | post-operative 1 month
  Assess adverse events and serious adverse events and patient safety
Complications | post-operative 3 months
  Assess adverse events and serious adverse events and patient safety
Complications | post-operative 6 months
  Assess adverse events and serious adverse events and patient safety
Complications | post-operative 12 months
  Assess adverse events and serious adverse events and patient safety
Incidence of cuff re-tears | post-operative 10 days
  Perform shoulder exam
Incidence of cuff re-tears | post-operative 3 months
  Perform shoulder exam and MRI to determine rate of re-tears
Incidence of cuff re-tears | post-operative 6 months
  Perform shoulder exam and MRI to determine rate of re-tears
Incidence of cuff re-tears | post-operative 12 months
  Perform shoulder exam and MRI to determine rate of re-tears

SECONDARY OUTCOMES:
Change from baseline Visual Analog Scale Score VAS | Baseline, Post-operative 10 days, and 1,3,6, and 12 months
  Assessment of patients shoulder pain 0-10, 10 being the worst
Change from baseline Euro Quality of Life five questionnaire EQ-5D-5L | Baseline, post-operative 3,6, and 12 months
  Assess the improvement of health in Mobility, Self care, Usual Activities, Pain/Discomfort., Anxiety/Depression and Overall health scale with 100 being the best
Change from baseline Constant-Mulrey Score | Baseline, post-operative 3,6, and 12 months
  The test is divided into four subscales: pain (15 points), activities of daily living (20 points), strength (25 points) and range of motion: forward elevation, external rotation, abduction and internal rotation of the shoulder (40 points). The higher the score, the higher the quality of the function.
Change from baseline Penn Shoulder Score | Baseline, post-operative 3,6, and 12 months
  Assessment of pain and satisfaction of should pain, This is a patient-reported outcome tool, and the scores range from 0 to 100 with a score of 100 indicating low pain, high satisfaction, and high function.
Western Ontario Rotator Cuff Index | Baseline, post-operative 3,6, and 12 months
  Assessment of symptoms, work, sports and recreational activities. Each question uses a visual analogue scale (VAS) - which is a straight line, representing a 100-point scale, ranging from 0-100. The maximum score is 2100 (worst possible symptoms). Zero (0) represents no symptoms at all.
Analysis of cuff integrity | Baseline, post-operative 3,6, and 12 months
  MRI Magnetic Resonance Imaging of shoulder to determine rate of re-tears

OTHER OUTCOMES:
Hematology testing Comprehensive Metabolic panel | Prior to surgery to confirm eligibility
  Measure many different components and characteristics of blood, which may include a red blood cell count, white blood cell count and/or the number of each type of white blood cells, platelet count, hemoglobin and hematocrit.
Whole blood and PRP (Plasma Rich Platelets) to be collected | Baseline, post-operative 3,6, and 12 months
  Change in baseline, A sample of whole blood and PRP will be transported to a central laboratory to perform cell and protein characterization to support exploratory outcomes.

CONTACTS AND LOCATIONS:
Locations (9):
- United States (9):
  - American Sports Medicine Institute, Birmingham, Alabama
  - Tucson Orthopedics, Tucson, Arizona
  - Holy Cross Orthopedic Research Institute, Fort Lauderdale, Florida
  - The Orthopaedic Research Foundation, Inc., Indianapolis, Indiana
  - Johns Hopkins University, Columbia, Maryland
  - University of Buffalo Orthopaedic & Sports Medicine, Buffalo, New York
  - Rothman Orthopaedic Institute, Philadelphia, Pennsylvania
  - University Orthopedics Center, State College, Pennsylvania
  - OrthoVirginia, Richmond, Virginia

IPD SHARING:
Plan to Share IPD: No